CLINICAL TRIAL: NCT04476732
Title: Interactions Between Skincare Product Ingredients and the Skin Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1529276
Record Dates: First submitted 2020-05-15; First posted 2020-07-20 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Dysbiosis
Keywords: microbiome; skincare; skin; paraben; phthalate
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paraben-free then Paraben-containing (Experimental): Paraben free facial lotion is applied twice a day for 1 week and measurements are taken. Then, paraben-containing facial lotion is applied twice a day for 1 week and measurements are taken.
  Interventions: Other: Paraben-free skincare product; Other: Paraben-containing skincare product

INTERVENTIONS:
Other: Paraben-free skincare product — Paraben-free lotion will be applied twice a day for one week.
Other: Paraben-containing skincare product — Paraben-containing lotion will be applied twice a day for one week.

SUMMARY:
This is a study of the influence of skincare products containing chemicals such as parabens and phthalates on the skin microbiome.

DETAILED DESCRIPTION:
Skin serves as a critical barrier between our bodies and the environment and the locus for a diverse and active microbial community. The composition and metabolic activity of the microbial community on the skin is presumably influenced by the local chemical environment, which includes natural skin lipids (e.g., squalene and sapienic acid), components of personal care products applied directly to skin, and semi-volatile organic compounds (SVOCs) that reach the skin through gas phase absorption, dust deposition, and direct contact with surfaces. Common semi-volatile ingredients in skin care products include phthalates, parabens, and UV blocking compounds (e.g., oxybenzone, octocrylene or homosalate).

The investigators have recently demonstrated a method of collecting chemicals from areas of skin with infrequent direct dermal contact using alcohol wipes to assess passive air to skin partitioning of both target and nontarget compounds (Garrido et al., in review). Low-volatility reaction products can accumulate in skin oils and act as skin irritants, with the potential of being absorbed into the bloodstream. With methods developed for chemical and microbiome sampling, the overall goal of the proposed research is to develop an understanding of the two-way interaction between organic chemicals on the skin and the composition of the skin microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 15 and over
* No known medical conditions that, in the investigator's opinion, may interfere with study participation.

Exclusion Criteria:

* Individuals who have been on any medication (including antibiotics, probiotics, prebiotics) that has caused a change in current skin composition of interest based on the opinion of the investigator.
* Individuals with systemic antibiotic use within last 60 days.
* Individuals with topical antibiotic use on the test sites within last 30 days
* Individuals unwilling/unable to avoid topical antibiotics, systemic antibiotics, prebiotics, and probiotics during study.
* No other interfering skin products should be used during duration of study. (Paraben-free & phthalate-free personal product "safe" list will be provided for other uses during study period if needed).
* Individuals unwilling or unable to undergo 1 week wash-in with paraben/phthalate-free products if needed in the opinion of the investigator.
* Female volunteers who are pregnant or are actively breastfeeding or planning a pregnancy within two months. (There is no known concern for risk to fetus but pregnancy can alter the microbiome being studied)
* Female volunteers who have started a new hormonal birth control agent or switched to a hormonal birth control agent within the past 60 days
* Individuals using any interfering skin products in the opinion of the investigator within 2 weeks of enrollment into the study.
* Individuals who have participated in any other clinical studies using the same test sites (face) in the past 14 days
* Individuals with a known history of hypersensitivity to any ingredients to the cosmetic agent that is being assessed
* Individuals who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study at the discretion of the investigator.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Change in detected paraben levels | Baseline, 1 week, 2 weeks
  Demonstrate the ability to detect chemicals (specifically parabens) found in common ingredients in personal care products on human skin. Collection of isopropyl alcohol forehead wipe and subsequent detection and quantification of parabens by GC-QTOF-MS (gas chromatography) and LC-QTOF-MS (liquid chromatography). Comparisons between baseline, week 1, and week 2 will be made.

SECONDARY OUTCOMES:
Influence of skincare product ingredient (specifically parabens) on facial skin microbiome | Baseline, 1 week, 2 weeks
  Document changes in microbial community composition following application of skin care ingredients of controversial concern (parabens) in comparison with changes following application of products not containing these ingredients. This is assessed by facial swab collections, DNA extraction, and determination of a list of specific bacterial species present at each time point. Comparisons between baseline, week 1, and week 2 will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — UC Davis Dermatology Clinical Trials Unit
Locations (1):
- UC Davis Dermatology Department, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No